CLINICAL TRIAL: NCT00792909
Title: Vaccination Course in Children Primed and Boosted With Pneumococcal Vaccine GSK 1024850A and in Age-matched Unprimed Children
Brief Title: Vaccination Course in Primed Children and Age-matched Unprimed Children With Pneumococcal Vaccine GSK1024850A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111736
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-05

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal vaccine; Pneumococcal disease; Safety; Immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections

ARMS (3):
- Synflorix™ Group 1 (Experimental): Subjects previously vaccinated with the Synflorix™ vaccine according to a 2+1 schedule, receiving one dose of Synflorix™ at 36-46 months of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A
- Synflorix™ Group 2 (Experimental): Subjects previously vaccinated with the Synflorix™ vaccine according to a 3+1 schedule, receiving one dose of Synflorix™ at 36-46 months of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A
- Unprimed Group (Active Comparator): Age-matched subjects not previously vaccinated with any pneumococcal vaccine receiving two doses of Synflorix™ at 36-46 and 38-48 months of age. Age-matching was ensured by the enrolment of subjects 36-46 months of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A — Intramuscular injection, 1 dose
  Arms: Synflorix™ Group 1; Synflorix™ Group 2
Biological: Pneumococcal conjugate vaccine GSK1024850A — Intramuscular injection, 2 doses
  Arms: Unprimed Group

SUMMARY:
The purpose of this study is to assess the immune memory induced by primary and booster vaccination with pneumococcal conjugate vaccine GSK1024850A in the first year of life through evaluation of the immune responses following vaccination with a booster dose of pneumococcal conjugate vaccine GSK1024850A in the fourth year of life and to assess immune responses following vaccination with a single dose of pneumococcal conjugate vaccine GSK1024850A in age-matched unprimed children.

The study also aims to assess the antibody persistence in the fourth year of life following primary and booster vaccination with pneumococcal conjugate vaccine GSK1024850A in the first year of life.

The study is also designed to evaluate the immunogenicity in terms of antibody response and the safety/reactogenicity in terms of solicited and unsolicited symptoms and serious adverse events following a 2-dose vaccination with pneumococcal conjugate vaccine GSK1024850A in the fourth year of life.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = 00307034)

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, +- 36-46 months of age at the time of vaccination.
* For primed subjects: having completed the full vaccination course with GSK1024850A in the primary study (NCT00307034).
* Subjects for whom the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/guardian(s) of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of the study vaccines, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to vaccination.
* For primed subjects: administration of any pneumococcal vaccine since the end of the primary study (NCT00307034).
* For unprimed subjects: previous vaccination with any pneumococcal vaccine.
* Administration of immunoglobulins and/or any blood products less than 6 months prior to the vaccination or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of reactions or allergic disease likely to be exacerbated by any component of the study vaccine.
* Acute disease at the time of enrolment.

Ages: 36 Months to 46 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2008-12-02 (Actual); Primary Completion 2009-07-02 (Actual); Study Completion 2009-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Slovakia (3):
  - GSK Investigational Site, Dlhá nad Oravou
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Ružomberok
- Sweden (2):
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Silfverdal SA, Skerlikova H, Zanova M, Papuchova D, Traskine M, Borys D, Schuerman L. Anamnestic immune response in 3- to 4-year-old children previously immunized with 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine as 2-dose or 3-dose priming and a booster dose in the first year of life. Pediatr Infect Dis J. 2011 Sep;30(9):e155-63. doi: 10.1097/INF.0b013e31821feeb7. PMID 21572373
- [Background] Silfverdal SA et al. Assessment of immunological memory following PHiD-CV immunisation according to 2+1 or 3+1 schedules in the first year of life. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Silfverdal SA et al. Immunogenicity/reactogenicity of 2-dose catch-up vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein-D conjugate vaccine (PHiD-CV) during fourth year of life. Abstract presented at the 8th Biennial International Symposium on Pneumococci & Pneumococcal Diseases (ISPPD), Foz de Iguaçu, Brazil, 11-15 March 2012.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an extension study of study 10PN-PD-DIT-002 (105539) for the primed subjects, and a self-contained study for the unprimed subjects.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/ exclusion criteria, contraindications/ precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Synflorix™ Group 2: Subjects previously vaccinated with the Synflorix™ vaccine according to a 3+1 schedule, receiving one dose of Synflorix™ at 36-46 months of age,
Period: Overall Study
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2 | Unprimed Group
Started | 51 | 59 | 62
Completed | 51 | 58 | 62
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Synflorix™ Group 1: Subjects previously vaccinated with the C™ vaccine according to a 2+1 schedule, receiving one dose of Synflorix™ at 36-46 months of age.
- Total: Total of all reporting groups
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2 | Unprimed Group | Total
Number analyzed (Participants) | 51 | 59 | 62 | 172
Age, Continuous [Geometric Mean (Standard Deviation); unit: Months] | 38.2 (1.83) | 38.0 (1.81) | 40.1 (2.64) | 38.82 (2.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 31 | 81
  Male | 26 | 34 | 31 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European heritage | 50 | 59 | 59 | 168
  Asian - central/ south Asian heritage | 0 | 0 | 1 | 1
  Asian - east Asian heritage | 0 | 0 | 1 | 1
  Asian - south east Asian heritage | 0 | 0 | 1 | 1
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Unprimed Group
Description: Antibodies assessed were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) and were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration greater than or equal to (≥) 0.05 μg/mL.
Time Frame: Pre-vaccination (PRE/ Day 0)
Population: The According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects with available immunogenicity data. This included subjects for whom assay results were available for antibodies against at least one pneumococcal vaccine serotype or protein D after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
μg/mL
  Anti-1 at PRE | 0.06 [0.05 to 0.08]
  Anti-4 at PRE | 0.04 [0.03 to 0.05]
  Anti-5 at PRE | 0.07 [0.05 to 0.09]
  Anti-6B at PRE | 0.1 [0.07 to 0.13]
  Anti-7F at PRE | 0.08 [0.05 to 0.12]
  Anti-9V at PRE | 0.05 [0.04 to 0.07]
  Anti-14 at PRE | 0.25 [0.16 to 0.38]
  Anti-18C at PRE | 0.06 [0.04 to 0.08]
  Anti-19F at PRE | 0.23 [0.14 to 0.38]
  Anti-23F at PRE | 0.06 [0.04 to 0.08]

2. Primary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Unprimed Group
Description: Antibodies assessed were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) and were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: One week after dose 1 (Day 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
μg/mL
  Anti-1 at Day 7 | 0.6 [0.47 to 0.76]
  Anti-4 at Day 7 | 2.37 [1.91 to 2.94]
  Anti-5 at Day 7 | 0.45 [0.34 to 0.59]
  Anti-6B at Day 7: number analyzed (Participants) | 58
  Anti-6B at Day 7 | 0.2 [0.14 to 0.29]
  Anti-7F at Day 7 | 0.92 [0.67 to 1.25]
  Anti-9V at Day 7 | 0.33 [0.23 to 0.48]
  Anti-14 at Day 7 | 0.54 [0.34 to 0.86]
  Anti-18C at Day 7: number analyzed (Participants) | 59
  Anti-18C at Day 7 | 1.45 [1.01 to 2.06]
  Anti-19F at Day 7: number analyzed (Participants) | 59
  Anti-19F at Day 7 | 1.82 [1.27 to 2.6]
  Anti-23F at Day 7 | 0.1 [0.07 to 0.15]

3. Primary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Unprimed Group
Description: as for outcome 2
Time Frame: One month after dose 2 (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
μg/mL
  Anti-1 at Month 3 | 2.81 [2.25 to 3.51]
  Anti-4 at Month 3 | 8.44 [7.16 to 9.94]
  Anti-5 at Month 3 | 3.54 [2.96 to 4.23]
  Anti-6B at Month 3 | 1.11 [0.84 to 1.46]
  Anti-7F at Month 3 | 6.1 [4.99 to 7.46]
  Anti-9V at Month 3 | 2.22 [1.74 to 2.82]
  Anti-14 at Month 3 | 6.48 [4.98 to 8.44]
  Anti-18C at Month 3 | 22.28 [18.14 to 27.36]
  Anti-19F at Month 3 | 17.03 [13.38 to 21.68]
  Anti-23F at Month 3 | 1.09 [0.81 to 1.45]

4. Primary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Synflorix Group 1 and Synflorix Group 2
Description: as for outcome 2
Time Frame: 1 month after booster dose (Month 10) - in primary study (105539)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
μg/mL
  Anti-1 at Month 10 | 1.91 [1.52 to 2.42] | 1.87 [1.49 to 2.33]
  Anti-4 at Month 10 | 2.97 [2.34 to 3.77] | 3.2 [2.62 to 3.91]
  Anti-5 at Month 10 | 2.71 [2.15 to 3.41] | 3.01 [2.4 to 3.76]
  Anti-6B at Month 10 | 0.9 [0.59 to 1.36] | 1.62 [1.16 to 2.27]
  Anti-7F at Month 10 | 2.94 [2.4 to 3.59] | 3.88 [3.23 to 4.65]
  Anti-9V at Month 10 | 2.59 [2.03 to 3.31] | 3.81 [3.11 to 4.67]
  Anti-14 at Month 10 | 3.91 [3.05 to 5] | 5.22 [4.22 to 6.46]
  Anti-18C at Month 10 | 4.87 [3.77 to 6.29] | 5.52 [4.2 to 7.26]
  Anti-19F at Month 10 | 6.68 [5.2 to 8.59] | 6.6 [5.16 to 8.46]
  Anti-23F at Month 10 | 2.12 [1.52 to 2.97] | 2.67 [1.99 to 3.59]

5. Primary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Synflorix Group 1 and Synflorix Group 2
Description: as for outcome 2
Time Frame: Pre-additional dose at Month 34 in the current study (Month 34)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
μg/mL
  Anti-1 at Month 34: number analyzed (Participants) | 49 | 57
  Anti-1 at Month 34 | 0.13 [0.1 to 0.17] | 0.17 [0.14 to 0.22]
  Anti-4 at Month 34: number analyzed (Participants) | 48 | 54
  Anti-4 at Month 34 | 0.15 [0.1 to 0.23] | 0.19 [0.14 to 0.25]
  Anti-5 at Month 34 | 0.24 [0.19 to 0.31] | 0.33 [0.26 to 0.42]
  Anti-6B at Month 34: number analyzed (Participants) | 48 | 57
  Anti-6B at Month 34 | 0.5 [0.29 to 0.88] | 1.01 [0.62 to 1.64]
  Anti-7F at Month 34: number analyzed (Participants) | 49 | 56
  Anti-7F at Month 34 | 0.33 [0.24 to 0.46] | 0.51 [0.42 to 0.61]
  Anti-9V at Month 34 | 0.24 [0.18 to 0.33] | 0.49 [0.34 to 0.69]
  Anti-14 at Month 34: number analyzed (Participants) | 50 | 56
  Anti-14 at Month 34 | 0.62 [0.39 to 0.97] | 1.1 [0.69 to 1.75]
  Anti-18C at Month 34: number analyzed (Participants) | 50 | 56
  Anti-18C at Month 34 | 0.37 [0.26 to 0.54] | 0.49 [0.35 to 0.7]
  Anti-19F at Month 34: number analyzed (Participants) | 47 | 56
  Anti-19F at Month 34 | 1.42 [0.8 to 2.51] | 1.44 [0.82 to 2.53]
  Anti-23F at Month 34: number analyzed (Participants) | 49 | 56
  Anti-23F at Month 34 | 0.41 [0.23 to 0.71] | 0.67 [0.41 to 1.11]

6. Primary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Synflorix Group 1 and Synflorix Group 2
Description: as for outcome 2
Time Frame: One week after vaccination at Month 34+7 days (Mth34+D7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
μg/mL
  Anti-1 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-1 at Mth34+D7 | 4.06 [3.2 to 5.15] | 4.72 [3.77 to 5.92]
  Anti-4 at Mth34+D7: number analyzed (Participants) | 49 | 55
  Anti-4 at Mth34+D7 | 7.54 [5.98 to 9.5] | 9.97 [7.68 to 12.95]
  Anti-5 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-5 at Mth34+D7 | 5.38 [4.09 to 7.08] | 7.07 [5.51 to 9.09]
  Anti-6B at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-6B at Mth34+D7 | 4 [2.82 to 5.69] | 6.33 [4.75 to 8.45]
  Anti-7F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-7F at Mth34+D7 | 6.18 [5.05 to 7.56] | 7.27 [5.87 to 9.01]
  Anti-9V at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-9V at Mth34+D7 | 7.48 [5.88 to 9.51] | 10.17 [7.86 to 13.16]
  Anti-14 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-14 at Mth34+D7 | 13.42 [9.7 to 18.55] | 19.67 [14.97 to 25.84]
  Anti-18C at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-18C at Mth34+D7 | 17.12 [12.77 to 22.94] | 22.62 [17.58 to 29.11]
  Anti-19F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-19F at Mth34+D7 | 20.28 [15.71 to 26.19] | 30.55 [24.32 to 38.37]
  Anti-23F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-23F at Mth34+D7 | 6.23 [4.34 to 8.94] | 8.42 [6.38 to 11.11]

7. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations ≥ the Cut-off in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: as for outcome 2
Time Frame: 1 month after booster dose (Month 10) - in primary study (105539), pre-additional dose at Month 34 in the current study (Month 34) and one week after vaccination at Month 34+7 days (Mth34+ D7);
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
Participants
  Anti-1 at Month 10 | 50 | 57
  Anti-1 at Month 34: number analyzed (Participants) | 49 | 57
  Anti-1 at Month 34 | 43 | 55
  Anti-1 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-1 at Mth34+D7 | 50 | 55
  Anti-4 at Month 10 | 50 | 57
  Anti-4 at Month 34: number analyzed (Participants) | 48 | 54
  Anti-4 at Month 34 | 41 | 54
  Anti-4 at Mth34+D7: number analyzed (Participants) | 49 | 55
  Anti-4 at Mth34+D7 | 49 | 55
  Anti-5 at Month 10 | 50 | 57
  Anti-5 at Month 34 | 49 | 57
  Anti-5 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-5 at Mth34+D7 | 50 | 55
  Anti-6B at Month 10 | 45 | 54
  Anti-6B at Month 34: number analyzed (Participants) | 48 | 57
  Anti-6B at Month 34 | 43 | 56
  Anti-6B at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-6B at Mth34+D7 | 50 | 55
  Anti-7F at Month 10 | 50 | 57
  Anti-7F at Month 34: number analyzed (Participants) | 49 | 56
  Anti-7F at Month 34 | 47 | 56
  Anti-7F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-7F at Mth34+D7 | 50 | 55
  Anti-9V at Month 10 | 50 | 57
  Anti-9V at Month 34 | 48 | 56
  Anti-9V at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-9V at Mth34+D7 | 50 | 55
  Anti-14 at Month 10 | 50 | 57
  Anti-14 at Month 34: number analyzed (Participants) | 50 | 56
  Anti-14 at Month 34 | 50 | 56
  Anti-14 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-14 at Mth34+D7 | 50 | 55
  Anti-18C at Month 10 | 50 | 57
  Anti-18C at Month 34: number analyzed (Participants) | 50 | 56
  Anti-18C at Month 34 | 48 | 56
  Anti-18C at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-18C at Mth34+D7 | 50 | 55
  Anti-19F at Month 10 | 50 | 57
  Anti-19F at Month 34: number analyzed (Participants) | 47 | 56
  Anti-19F at Month 34 | 47 | 56
  Anti-19F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-19F at Mth34+D7 | 50 | 55
  Anti-23F at Month 10 | 49 | 56
  Anti-23F at Month 34: number analyzed (Participants) | 49 | 56
  Anti-23F at Month 34 | 43 | 56
  Anti-23F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-23F at Mth34+D7 | 49 | 55

8. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations ≥ the Cut-off in the Unprimed Group;
Description: as for outcome 2
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3);
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
Participants
  Anti-1 at PRE | 34
  Anti-1 at Day 7 | 60
  Anti-1 at Month 3 | 60
  Anti-4 at PRE | 9
  Anti-4 at Day 7 | 60
  Anti-4 at Month 3 | 60
  Anti-5 at PRE | 37
  Anti-5 at Day 7 | 60
  Anti-5 at Month 3 | 60
  Anti-6B at PRE | 40
  Anti-6B at Day 7: number analyzed (Participants) | 58
  Anti-6B at Day 7 | 49
  Anti-6B at Month 3 | 60
  Anti-7F at PRE | 29
  Anti-7F at Day 7 | 60
  Anti-7F at Month 3 | 60
  Anti-9V at PRE | 21
  Anti-9V at Day 7 | 58
  Anti-9V at Month 3 | 60
  Anti-14 at PRE | 56
  Anti-14 at Day 7 | 58
  Anti-14 at Month 3 | 60
  Anti-18C at PRE | 23
  Anti-18C at Day 7: number analyzed (Participants) | 59
  Anti-18C at Day 7 | 59
  Anti-18C at Month 3 | 60
  Anti-19F at PRE | 44
  Anti-19F at Day 7: number analyzed (Participants) | 59
  Anti-19F at Day 7 | 59
  Anti-19F at Month 3 | 60
  Anti-23F at PRE | 23
  Anti-23F at Day 7 | 39
  Anti-23F at Month 3 | 60

9. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations ≥ the Cut-off in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.2 μg/mL.
Time Frame: 1 month after booster dose (Month 10) - in primary study (105539), pre-additional dose at Month 34 in the current study (Month 34) and one week after vaccination at Month 34+7 days (Mth34+D7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
Participants
  Anti-1 at Month 10 | 50 | 57
  Anti-1 at Month 34: number analyzed (Participants) | 49 | 57
  Anti-1 at Month 34 | 16 | 28
  Anti-1 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-1 at Mth34+D7 | 50 | 55
  Anti-4 at Month 10 | 50 | 57
  Anti-4 at Month 34: number analyzed (Participants) | 48 | 54
  Anti-4 at Month 34 | 12 | 20
  Anti-4 at Mth34+D7: number analyzed (Participants) | 49 | 55
  Anti-4 at Mth34+D7 | 49 | 55
  Anti-5 at Month 10 | 50 | 57
  Anti-5 at Month 34 | 31 | 35
  Anti-5 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-5 at Mth34+D7 | 50 | 55
  Anti-6B at Month 10 | 44 | 54
  Anti-6B at Month 34: number analyzed (Participants) | 48 | 57
  Anti-6B at Month 34 | 29 | 44
  Anti-6B at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-6B at Mth34+D7 | 49 | 55
  Anti-7F at Month 10 | 50 | 57
  Anti-7F at Month 34: number analyzed (Participants) | 49 | 56
  Anti-7F at Month 34 | 37 | 53
  Anti-7F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-7F at Mth34+D7 | 50 | 55
  Anti-9V at Month 10 | 49 | 57
  Anti-9V at Month 34 | 27 | 45
  Anti-9V at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-9V at Mth34+D7 | 50 | 55
  Anti-14 at Month 10 | 50 | 57
  Anti-14 at Month 34: number analyzed (Participants) | 50 | 56
  Anti-14 at Month 34 | 37 | 49
  Anti-14 at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-14 at Mth34+D7 | 50 | 55
  Anti-18C at Month 10 | 50 | 56
  Anti-18C at Month 34: number analyzed (Participants) | 50 | 56
  Anti-18C at Month 34 | 35 | 44
  Anti-18C at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-18C at Mth34+D7 | 50 | 55
  Anti-19F at Month 10 | 49 | 56
  Anti-19F at Month 34: number analyzed (Participants) | 47 | 56
  Anti-19F at Month 34 | 39 | 47
  Anti-19F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-19F at Mth34+D7 | 50 | 55
  Anti-23F at Month 10 | 47 | 55
  Anti-23F at Month 34: number analyzed (Participants) | 49 | 56
  Anti-23F at Month 34 | 29 | 36
  Anti-23F at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-23F at Mth34+D7 | 49 | 55

10. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations ≥ the Cut-off in the Unprimed Group
Description: Antibodies assessed were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C,19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) and were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.20 μg/mL.
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3);
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
Participants
  Anti-1 at PRE | 10
  Anti-1 at Day 7 | 54
  Anti-1 at Month 3 | 60
  Anti-4 at PRE | 4
  Anti-4 at Day 7 | 60
  Anti-4 at Month 3 | 60
  Anti-5 at PRE | 9
  Anti-5 at Day 7 | 47
  Anti-5 at Month 3 | 60
  Anti-6B at PRE | 19
  Anti-6B at Day 7: number analyzed (Participants) | 58
  Anti-6B at Day 7 | 29
  Anti-6B at Month 3 | 56
  Anti-7F at PRE | 11
  Anti-7F at Day 7 | 54
  Anti-7F at Month 3 | 60
  Anti-9V at PRE | 7
  Anti-9V at Day 7 | 40
  Anti-9V at Month 3 | 60
  Anti-14 at PRE | 27
  Anti-14 at Day 7 | 42
  Anti-14 at Month 3 | 60
  Anti-18C at PRE | 8
  Anti-18C at Day 7: number analyzed (Participants) | 59
  Anti-18C at Day 7 | 56
  Anti-18C at Month 3 | 60
  Anti-19F at PRE | 29
  Anti-19F at Day 7: number analyzed (Participants) | 59
  Anti-19F at Day 7 | 57
  Anti-19F at Month 3 | 60
  Anti-23F at PRE | 11
  Anti-23F at Day 7 | 16
  Anti-23F at Month 3 | 56

11. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: Seropositivity status was defined as opsonophacocytic activity against pneumococcal serotypes ≥ 8.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 48 | 55
Titers
  Opsono-1 at Month 10: number analyzed (Participants) | 44 | 53
  Opsono-1 at Month 10 | 243.9 [137.3 to 433.3] | 176.9 [104 to 301]
  Opsono-1 at Month 34: number analyzed (Participants) | 47 | 55
  Opsono-1 at Month 34 | 5.5 [4.3 to 7] | 6.2 [4.9 to 8]
  Opsono-1 at Mth34+D7 | 2342.2 [1788.8 to 3066.7] | 2321.5 [1827.1 to 2949.7]
  Opsono-4 at Month 10: number analyzed (Participants) | 43 | 55
  Opsono-4 at Month 10 | 937.6 [600.8 to 1463.4] | 1347 [1068.8 to 1697.7]
  Opsono-4 at Month 34: number analyzed (Participants) | 44 | 52
  Opsono-4 at Month 34 | 9.6 [4.9 to 18.8] | 9.5 [5.8 to 15.6]
  Opsono-4 at Mth34+D7: number analyzed (Participants) | 48 | 53
  Opsono-4 at Mth34+D7 | 13247.5 [9898 to 17730.4] | 17732.6 [13218.8 to 23787.7]
  Opsono-5 at Month 10: number analyzed (Participants) | 45 | 54
  Opsono-5 at Month 10 | 154 [94.2 to 251.6] | 181.2 [125.4 to 262]
  Opsono-5 at Month 34: number analyzed (Participants) | 47 | 54
  Opsono-5 at Month 34 | 6.7 [5.2 to 8.6] | 8 [6.1 to 10.6]
  Opsono-5 at Mth34+D7 | 991.5 [769.8 to 1277.1] | 1221.1 [912.4 to 1634.2]
  Opsono-6B at Month 10: number analyzed (Participants) | 44 | 51
  Opsono-6B at Month 10 | 292.2 [147.1 to 580.3] | 458.8 [254.8 to 825.9]
  Opsono-6B at Month 34: number analyzed (Participants) | 42 | 54
  Opsono-6B at Month 34 | 61.5 [22.8 to 165.6] | 126.3 [59.4 to 268.5]
  Opsono-6B at Mth34+D7: number analyzed (Participants) | 47 | 54
  Opsono-6B at Mth34+D7 | 3312.9 [1751.2 to 6267.2] | 3136 [1730 to 5684.6]
  Opsono-7F at Month 10: number analyzed (Participants) | 44 | 53
  Opsono-7F at Month 10 | 2257.8 [1601.9 to 3182.3] | 3856.8 [2890.4 to 5146.2]
  Opsono-7F at Month 34: number analyzed (Participants) | 45 | 53
  Opsono-7F at Month 34 | 1329.1 [778.8 to 2268.4] | 1225.5 [842.5 to 1782.6]
  Opsono-7F at Mth34+D7: number analyzed (Participants) | 48 | 52
  Opsono-7F at Mth34+D7 | 20779 [14616.7 to 29539.1] | 22461.4 [16876.9 to 29893.7]
  Opsono-9V at Month 10: number analyzed (Participants) | 44 | 54
  Opsono-9V at Month 10 | 1581.7 [1147.7 to 2179.9] | 2013.9 [1565.3 to 2591]
  Opsono-9V at Month 34: number analyzed (Participants) | 43 | 53
  Opsono-9V at Month 34 | 307.4 [210.3 to 449.4] | 292.3 [221 to 386.6]
  Opsono-9V at Mth34+D7: number analyzed (Participants) | 48 | 52
  Opsono-9V at Mth34+D7 | 21193.6 [16100.3 to 27898.2] | 19038.4 [14154.7 to 25607.2]
  Opsono-14 at Month 10: number analyzed (Participants) | 35 | 52
  Opsono-14 at Month 10 | 1092.5 [691.9 to 1725] | 1207.1 [961.4 to 1515.5]
  Opsono-14 at Month 34: number analyzed (Participants) | 41 | 49
  Opsono-14 at Month 34 | 421.5 [258.8 to 686.5] | 738.6 [540 to 1010.2]
  Opsono-14 at Mth34+D7: number analyzed (Participants) | 48 | 54
  Opsono-14 at Mth34+D7 | 14310 [10214 to 20048.7] | 14670.9 [10258 to 20982.2]
  Opsono-18C at Month 10: number analyzed (Participants) | 45 | 54
  Opsono-18C at Month 10 | 375.8 [251.3 to 562.1] | 567.4 [422.8 to 761.5]
  Opsono-18C at Month 34: number analyzed (Participants) | 45 | 54
  Opsono-18C at Month 34 | 11 [6 to 20.2] | 17.7 [9.6 to 32.9]
  Opsono-18C at Mth34+D7: number analyzed (Participants) | 48 | 51
  Opsono-18C at Mth34+D7 | 6095.8 [4090.7 to 9083.8] | 6448.7 [4258.7 to 9764.9]
  Opsono-19F at Month 10: number analyzed (Participants) | 43 | 54
  Opsono-19F at Month 10 | 463.7 [318.3 to 675.6] | 950.5 [653.3 to 1383]
  Opsono-19F at Month 34: number analyzed (Participants) | 47 | 55
  Opsono-19F at Month 34 | 34.1 [18.4 to 63.2] | 48.4 [25.9 to 90.6]
  Opsono-19F at Mth34+D7 | 2231.5 [1267.7 to 3927.9] | 5684.4 [3647.8 to 8858]
  Opsono-23F at Month 10: number analyzed (Participants) | 45 | 53
  Opsono-23F at Month 10 | 1414.6 [827.9 to 2417.1] | 1984.8 [1520.3 to 2591.3]
  Opsono-23F at Month 34: number analyzed (Participants) | 43 | 49
  Opsono-23F at Month 34 | 458.5 [186.3 to 1128.2] | 465.6 [209.6 to 1034]
  Opsono-23F at Mth34+D7: number analyzed (Participants) | 48 | 54
  Opsono-23F at Mth34+D7 | 15688.3 [10571.2 to 23282.4] | 13812.6 [9566 to 19944.4]

12. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F in the Unprimed Group
Description: Seropositivity status was defined as opsonophacocytic activity against pneumococcal serotypes ≥ 8.
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Unprimed Group
Number analyzed (Participants) | 59
Titers
  Opsono-1 at PRE: number analyzed (Participants) | 58
  Opsono-1 at PRE | 4 [4 to 4]
  Opsono-1 at Day 7: number analyzed (Participants) | 58
  Opsono-1 at Day 7 | 441.1 [302.4 to 643.4]
  Opsono-1 at Month 3: number analyzed (Participants) | 56
  Opsono-1 at Month 3 | 103 [67.6 to 157]
  Opsono-4 at PRE: number analyzed (Participants) | 58
  Opsono-4 at PRE | 5.1 [3.9 to 6.7]
  Opsono-4 at Day 7: number analyzed (Participants) | 58
  Opsono-4 at Day 7 | 9675.9 [7792.2 to 12014.9]
  Opsono-4 at Month 3: number analyzed (Participants) | 56
  Opsono-4 at Month 3 | 2687.5 [2165 to 3336.1]
  Opsono-5 at PRE | 4.1 [3.9 to 4.5]
  Opsono-5 at Day 7: number analyzed (Participants) | 57
  Opsono-5 at Day 7 | 330 [200.5 to 543]
  Opsono-5 at Month 3: number analyzed (Participants) | 56
  Opsono-5 at Month 3 | 127.6 [92.7 to 175.6]
  Opsono-6B at PRE: number analyzed (Participants) | 55
  Opsono-6B at PRE | 21.6 [11 to 42.4]
  Opsono-6B at Day 7: number analyzed (Participants) | 54
  Opsono-6B at Day 7 | 438.2 [208.4 to 921.5]
  Opsono-6B at Month 3: number analyzed (Participants) | 57
  Opsono-6B at Month 3 | 1040.9 [652.8 to 1659.5]
  Opsono-7F at PRE: number analyzed (Participants) | 55
  Opsono-7F at PRE | 644.2 [355.5 to 1167.3]
  Opsono-7F at Day 7: number analyzed (Participants) | 57
  Opsono-7F at Day 7 | 11048.4 [8626.3 to 14150.5]
  Opsono-7F at Month 3: number analyzed (Participants) | 55
  Opsono-7F at Month 3 | 6213.1 [4793.1 to 8053.7]
  Opsono-9V at PRE: number analyzed (Participants) | 55
  Opsono-9V at PRE | 103.1 [53.8 to 197.6]
  Opsono-9V at Day 7: number analyzed (Participants) | 57
  Opsono-9V at Day 7 | 12217.8 [9359.1 to 15949.8]
  Opsono-9V at Month 3: number analyzed (Participants) | 55
  Opsono-9V at Month 3 | 6085.2 [4718.5 to 7847.9]
  Opsono-14 at PRE: number analyzed (Participants) | 55
  Opsono-14 at PRE | 252.5 [138.1 to 461.5]
  Opsono-14 at Day 7: number analyzed (Participants) | 57
  Opsono-14 at Day 7 | 3948.7 [2958.9 to 5269.5]
  Opsono-14 at Month 3: number analyzed (Participants) | 55
  Opsono-14 at Month 3 | 4978.9 [3857.8 to 6425.9]
  Opsono-18C at PRE: number analyzed (Participants) | 53
  Opsono-18C at PRE | 6.1 [4 to 9.3]
  Opsono-18C at Day 7: number analyzed (Participants) | 57
  Opsono-18C at Day 7 | 3905.6 [2648 to 5760.4]
  Opsono-18C at Month 3: number analyzed (Participants) | 56
  Opsono-18C at Month 3 | 3984.5 [3187.9 to 4980.2]
  Opsono-19F at PRE: number analyzed (Participants) | 48
  Opsono-19F at PRE | 8.4 [5.6 to 12.7]
  Opsono-19F at Day 7: number analyzed (Participants) | 57
  Opsono-19F at Day 7 | 367.5 [202.7 to 666.5]
  Opsono-19F at Month 3: number analyzed (Participants) | 56
  Opsono-19F at Month 3 | 1772.5 [1285.9 to 2443.3]
  Opsono-23F at PRE: number analyzed (Participants) | 52
  Opsono-23F at PRE | 265.3 [121.5 to 579.6]
  Opsono-23F at Day 7: number analyzed (Participants) | 58
  Opsono-23F at Day 7 | 5059 [3800.6 to 6734]
  Opsono-23F at Month 3: number analyzed (Participants) | 57
  Opsono-23F at Month 3 | 5095.5 [3992.3 to 6503.6]

13. Secondary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 6A and 19A in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: Antibodies assessed were those against the vaccine pneumococcal serotypes 6A and19A (ANTI-6A and19A) and were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
μg/mL
  Anti-6A at Month 10: number analyzed (Participants) | 49 | 57
  Anti-6A at Month 10 | 0.31 [0.2 to 0.48] | 0.51 [0.33 to 0.77]
  Anti-6A at Month 34: number analyzed (Participants) | 48 | 55
  Anti-6A at Month 34 | 0.26 [0.16 to 0.42] | 0.45 [0.28 to 0.71]
  Anti-6A at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-6A at Mth34+D7 | 1.13 [0.71 to 1.79] | 2 [1.32 to 3.03]
  Anti-19A at Month 10 | 0.8 [0.53 to 1.2] | 0.75 [0.5 to 1.12]
  Anti-19A at Month 34: number analyzed (Participants) | 49 | 57
  Anti-19A at Month 34 | 0.31 [0.2 to 0.49] | 0.26 [0.17 to 0.4]
  Anti-19A at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-19A at Mth34+D7 | 3.44 [2.3 to 5.15] | 3.76 [2.47 to 5.73]

14. Secondary Outcome: Antibody Geometric Mean Concentrations (GMCs) Against the Vaccine Pneumococcal Serotypes 6A and 19A in the Unprimed Group
Description: Antibodies assessed were those against the vaccine pneumococcal serotypes 6A and 19A (ANTI-6A and 19A) and were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
μg/mL
  Anti-6A at PRE | 0.11 [0.08 to 0.16]
  Anti-6A at Day 7 | 0.15 [0.11 to 0.21]
  Anti-6A at Month 3 | 0.58 [0.42 to 0.79]
  Anti-19A at PRE | 0.13 [0.09 to 0.2]
  Anti-19A at Day 7: number analyzed (Participants) | 59
  Anti-19A at Day 7 | 0.32 [0.21 to 0.49]
  Anti-19A at Month 3 | 1.97 [1.46 to 2.65]

15. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 6A and 19A Antibody Concentrations ≥ the Cut-off in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: as for outcome 14
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
Participants
  Anti-6A at Month 10: number analyzed (Participants) | 49 | 57
  Anti-6A at Month 10 | 42 | 51
  Anti-6A at Month 34: number analyzed (Participants) | 48 | 55
  Anti-6A at Month 34 | 43 | 51
  Anti-6A at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-6A at Mth34+D7 | 48 | 55
  Anti-19A at Month 10 | 48 | 54
  Anti-19A at Month 34: number analyzed (Participants) | 49 | 57
  Anti-19A at Month 34 | 44 | 50
  Anti-19A at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-19A at Mth34+D7 | 50 | 55

16. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 6A and 19A Antibody Concentrations ≥ the Cut-off in the Unprimed Group
Description: as for outcome 14
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
Participants
  Anti-6A at PRE | 47
  Anti-6A at Day 7 | 50
  Anti-6A at Month 3 | 59
  Anti-19A at PRE | 41
  Anti-19A at Day 7: number analyzed (Participants) | 59
  Anti-19A at Day 7 | 55
  Anti-19A at Month 3 | 60

17. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 6A and 19A Antibody Concentrations ≥ the Cut-off in the Synflorix™ Group 1 and Synflorix™ Group 2;
Description: Antibodies assessed were those against the vaccine pneumococcal serotypes 6A and 19A (ANTI-6A and 19A) and were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (μg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.20 μg/mL.
Time Frame: 1 month after booster dose (Month 10) - in primary study (105539), pre-additional dose at Month 34 in the current study (Month 34) and one week after vaccination at Month 34+7 days (Mth34+D7);
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
Participants
  Anti-6A at Month 10: number analyzed (Participants) | 49 | 57
  Anti-6A at Month 10 | 31 | 43
  Anti-6A at Month 34: number analyzed (Participants) | 48 | 55
  Anti-6A at Month 34 | 22 | 38
  Anti-6A at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-6A at Mth34+D7 | 44 | 51
  Anti-19A at Month 10 | 41 | 45
  Anti-19A at Month 34: number analyzed (Participants) | 49 | 57
  Anti-19A at Month 34 | 26 | 30
  Anti-19A at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-19A at Mth34+D7 | 47 | 54

18. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 6A and 19A Antibody Concentrations ≥ 0.20 μg/mL in the Unprimed Group
Description: as for outcome 17
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
Participants
  Anti-6A at PRE | 13
  Anti-6A at Day 7 | 24
  Anti-6A at Month 3 | 49
  Anti-19A at PRE | 22
  Anti-19A at Day 7: number analyzed (Participants) | 59
  Anti-19A at Day 7 | 33
  Anti-19A at Month 3 | 58

19. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 6A and 19A in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: Seropositivity status defined as opsonophacocytic activity against pneumococcal serotypes ≥ 8
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 48 | 55
Titers
  Opsono-6A at Month 10: number analyzed (Participants) | 35 | 44
  Opsono-6A at Month 10 | 60.9 [25.9 to 143.1] | 135 [68.3 to 267]
  Opsono-6A at Month 34: number analyzed (Participants) | 40 | 47
  Opsono-6A at Month 34 | 64.3 [27.1 to 152.7] | 81.5 [39.7 to 167.5]
  Opsono-6A at Mth34+D7: number analyzed (Participants) | 45 | 50
  Opsono-6A at Mth34+D7 | 1639.4 [958.6 to 2803.9] | 1267.3 [713.8 to 2250]
  Opsono-19A at Month 10: number analyzed (Participants) | 36 | 46
  Opsono-19A at Month 10 | 14.4 [7.6 to 27.3] | 35.9 [18 to 71.6]
  Opsono-19A at Month 34: number analyzed (Participants) | 45 | 55
  Opsono-19A at Month 34 | 8 [5.2 to 12.2] | 8.6 [5.6 to 13.4]
  Opsono-19A at Mth34+D7 | 799.3 [372.8 to 1713.4] | 1871.6 [975.8 to 3589.8]

20. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes 6A and 19A in the Unprimed Group
Description: Seropositivity status defined as opsonophacocytic activity against pneumococcal serotypes ≥ 8.
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Unprimed Group
Number analyzed (Participants) | 58
Titers
  Opsono-6A at PRE: number analyzed (Participants) | 50
  Opsono-6A at PRE | 36.3 [18.9 to 69.6]
  Opsono-6A at Day: number analyzed (Participants) | 52
  Opsono-6A at Day | 389.6 [215.2 to 705.5]
  Opsono-6A at Month: number analyzed (Participants) | 52
  Opsono-6A at Month | 715.2 [487.3 to 1049.6]
  Opsono-19A at PRE | 5.4 [4.2 to 6.9]
  Opsono-19A at Day 7: number analyzed (Participants) | 55
  Opsono-19A at Day 7 | 211.9 [99.9 to 449.7]
  Opsono-19A at Month 3: number analyzed (Participants) | 53
  Opsono-19A at Month 3 | 406.4 [227.3 to 726.9]

21. Secondary Outcome: Concentrations of Antibodies Against Protein D (ANTI-PD) in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: ANTI-PD concentrations were expressed as geometric mean concentrations (GMCs), in enzyme-linked immunosorbent assay (ELISA) unit per milliliter (EL.U/mL). Seropositivity status was defined as Anti-PD antibody concentrations ≥ 100 EL.U/mL.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 50 | 57
EL.U/mL
  Anti-PD at Month 10: number analyzed (Participants) | 48 | 56
  Anti-PD at Month 10 | 1438 [1018.9 to 2029.4] | 2241.3 [1752.5 to 2866.3]
  Anti-PD at Month 34 | 301.6 [219.5 to 414.3] | 461.3 [351.1 to 606]
  Anti-PD at Mth34+D7: number analyzed (Participants) | 50 | 55
  Anti-PD at Mth34+D7 | 1724.1 [1299.4 to 2287.5] | 2113.2 [1651.2 to 2704.5]

22. Secondary Outcome: Concentrations of Antibodies Against Protein D (ANTI-PD) in the Unprimed Group
Description: as for outcome 21
Time Frame: Pre-vaccination (PRE/ Day 0), one week after dose 1 (Day 7) and one month after dose 2 (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Unprimed Group
Number analyzed (Participants) | 60
EL.U/mL
  Anti-PD at PRE | 110.9 [88.8 to 138.6]
  Anti-PD at Day 7 | 536.3 [390.7 to 736.2]
  Anti-PD at Month 3 | 960.4 [752.7 to 1225.5]

23. Secondary Outcome: Number of Subjects With B-cells Detection in the Synflorix™ Group 1 and Synflorix™ Group 2
Description: Quantification of memory B-cells that produce antibodies against vaccine pneumococcal serotypes (PS) 6B, 18C, 19F, 23F and C-PS (Elispot assay), prior to and 7-10 days post- additional dose.
Time Frame: Pre-additional dose at Month 34 in the current study (Month 34) and one week after vaccination at Month 34+7 days (Mth34+D7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2
Number analyzed (Participants) | 10 | 13
Participants
  18C PS at Month 34: number analyzed (Participants) | 10 | 11
  18C PS at Month 34 | 377 (459.3) | 424.9 (668.2)
  18C PS at Mth34+D7: number analyzed (Participants) | 7 | 13
  18C PS at Mth34+D7 | 1205.3 (661.4) | 2891.2 (2274.5)
  19F PS at Month 34: number analyzed (Participants) | 10 | 11
  19F PS at Month 34 | 163.1 (306.4) | 635.4 (1196.6)
  19F PS at Mth34+D7: number analyzed (Participants) | 7 | 13
  19F PS at Mth34+D7 | 856.7 (1211.7) | 1626 (1760.5)
  23F PS at Month 34: number analyzed (Participants) | 10 | 11
  23F PS at Month 34 | 174.2 (285) | 212.2 (320.8)
  23F PS at Mth34+D7: number analyzed (Participants) | 7 | 13
  23F PS at Mth34+D7 | 120.1 (92) | 351.9 (400.4)
  6B PS at Month 34: number analyzed (Participants) | 10 | 11
  6B PS at Month 34 | 136.1 (131.8) | 508.5 (606.3)
  6B PS at Mth34+D7: number analyzed (Participants) | 7 | 13
  6B PS at Mth34+D7 | 153.1 (216) | 469.7 (554.5)
  C-PS at Month 34: number analyzed (Participants) | 10 | 11
  C-PS at Month 34 | 246.3 (247.3) | 751.2 (790.5)
  C-PS at Mth34+D7: number analyzed (Participants) | 7 | 13
  C-PS at Mth34+D7 | 167.6 (92) | 600.5 (488.8)

24. Secondary Outcome: Number of Subjects With B-cells Detection in the Unprimed Group
Description: Quantification of memory B-cells that produce antibodies against vaccine pneumococcal serotypes (PS) 6B, 18C, 19F, 23F and C-PS (Elispot assay), prior to, and 7-10 days post-dose 1.
Time Frame: Pre-vaccination (PRE/ Day 0) and one week after dose 1 (Day 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Participants
Arm/Group | Unprimed Group
Number analyzed (Participants) | 13
Participants
  18C PS at PRE: number analyzed (Participants) | 12
  18C PS at PRE | 246.5 (310.8)
  18C PS at Day 7 | 3014.2 (4168.4)
  19F PS at PRE: number analyzed (Participants) | 12
  19F PS at PRE | 306.4 (423.1)
  19F PS at Day 7 | 599.8 (643.8)
  23F PS at PRE: number analyzed (Participants) | 12
  23F PS at PRE | 280 (492.2)
  23F PS at Day 7 | 450 (529.4)
  6B PS at PRE: number analyzed (Participants) | 12
  6B PS at PRE | 159.8 (220.7)
  6B PS at Day 7 | 432.4 (478.3)
  C-PS at PRE: number analyzed (Participants) | 12
  C-PS at PRE | 751.9 (463)
  C-PS at Day 7 | 789.2 (751.1)

25. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed local symptoms were pain, redness and swelling. Any = occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = crying when limb was moved/ spontaneously painful. Grade 3 Redness/ Swelling = Redness/ swelling at injection site greater than (>) 30 millimeters (mm).
Time Frame: During the 4-day (Days 0-3) post-vaccination period with the Synflorix™ vaccine, following the additional dose in the Synflorix Group1 and the Synflorix Group2 and across the 2 doses in the Unprimed Group
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2 | Unprimed Group
Number analyzed (Participants) | 51 | 59 | 62
Participants
  Any Pain | 41 | 44 | 49
  Grade 3 Pain | 3 | 4 | 6
  Any Redness | 34 | 35 | 41
  Grade 3 Redness | 9 | 12 | 15
  Any Swelling | 28 | 27 | 30
  Grade 3 Swelling | 5 | 9 | 9

26. Secondary Outcome: Number/ Percentage of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability/ fussiness (Irr./Fuss.), loss of appetite (Loss Appet.) and Fever (rectal temperature ≥ 38.0 °C). Any = occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Related = occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 drowsiness = drowsiness that prevented normal everyday activities. Grade 3 Irr./Fuss. = crying that could not be comforted/ prevented normal everyday activities. Grade 3 loss of appetite = not eating at all. Grade 3 fever = rectal temperature > 40.0°C.
Time Frame: During the 4-day (Days 0-3) post-vaccination period with the Synflorix™ vaccine, following the additional dose in the Synflorix Group 1 and the Synflorix Group 2 and across the 2 doses in the Unprimed Group.
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2 | Unprimed Group
Number analyzed (Participants) | 51 | 59 | 62
Participants
  Any Drowsiness | 20 | 23 | 17
  Grade 3 Drowsiness | 0 | 0 | 0
  Related Drowsiness | 20 | 23 | 17
  Any Fever | 9 | 5 | 8
  Grade 3 Fever | 0 | 0 | 0
  Related Fever | 9 | 4 | 7
  Any Irr./Fuss. | 20 | 27 | 21
  Grade 3 Irr./Fuss. | 0 | 0 | 0
  Related Irr./Fuss. | 20 | 25 | 20
  Any Loss Appet. | 12 | 13 | 14
  Grade 3 Loss Appet. | 0 | 0 | 0
  Related Loss Appet. | 12 | 13 | 14

27. Secondary Outcome: Number (%) of Subjects With Unsolicited Adverse Events
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any = occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination.
Time Frame: Within the 31-day (Days 0-30) period post vaccination, with the Synflorix™ vaccine, following the additional dose in the Synflorix group1 and the Synflorix Group 2 and across the 2 doses in the Unprimed Group
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2 | Unprimed Group
Number analyzed (Participants) | 51 | 59 | 62
Participants | 24 | 24 | 40

28. Secondary Outcome: Number (%) of Subjects With Serious Adverse Events
Description: A serious adverse event (SAE) was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalisation, as per the medical or scientific judgement of the physician. Any = occurrence of a SAE, regardless of relationship to vaccination.
Time Frame: During the 31-day period following vaccination period
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2 | Unprimed Group
Number analyzed (Participants) | 51 | 59 | 62
Participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms during the 4-day post-vaccination period and unsolicited AEs and SAEs: during the 31-day post-vaccination period, following additional dose in the Synflorix Group 1 and the Synflorix Group 2 and across the 2 doses in the Unprimed Group.
Arm/Group | Synflorix™ Group 1 | Synflorix™ Group 2 | Unprimed Group
All-Cause Mortality (participants affected / at risk) | 1/51 | 1/59 | 1/62
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/59 | 1/62
Other Adverse Events (participants affected / at risk) | 41/51 | 44/59 | 49/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix™ Group 1 (N=51) | Synflorix™ Group 2 (N=59) | Unprimed Group (N=62)
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix™ Group 1 (N=51) | Synflorix™ Group 2 (N=59) | Unprimed Group (N=62)
Bronchitis (Infections and infestations) | 2 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5
Irritability (Psychiatric disorders) | 20 | 27 | 21
Nasopharyngitis (Infections and infestations) | 1 | 4 | 12
Pain (General disorders) | 41 | 44 | 49
Pyrexia (General disorders) | 7 | 8 | 7
Swelling (General disorders) | 28 | 27 | 30
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 4
Viral infection (Infections and infestations) | 0 | 1 | 6
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2
Redness (General disorders) | 34 | 35 | 41
Drowsiness (General disorders) | 20 | 23 | 17
Fever (Rectally, ≥ 38.0°C) (General disorders) | 9 | 5 | 8
Loss of appetite (General disorders) | 12 | 13 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.